CLINICAL TRIAL: NCT07200141
Title: Simultaneous Boost in Neoadjuvant Radiotherapy for Rectal Cancer：A Phase 2, Randomized Controlled Study
Brief Title: Simultaneous Boost in Neoadjuvant Radiotherapy for Rectal Cancer
Acronym: SIB-NCRT-pumch
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: I-25PJ2066
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Rectal Adenocarcinoma
Keywords: locally advanced rectal cancer; Neoadjuvant Chemoradiotherapy; Dose Escalation; Simultaneous Integrated Boost
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (GTV 58.75 Gy/25f) (Experimental): Radiotherapy: long course simultaneous integrated boost radiotherapy
  * Gross tumor volume (GTV): A total dose of 58.75Gy delivered in 25 fractions using a simultaneous integrated boost approach.
  * CTV: 45Gy/25f
  * Mesorectum lymph node(GTVnd1):58.75Gy/25f
  * Lateral lymph node（GTVnd2）：60Gy/25f Concurrent Chemotherapy: Concurrent administration of capecitabine (825 mg/m² twice daily, 5 days per week) or XELOX regimen during radiotherapy After treatment, patients will undergo restaging and proceed to total mesorectal excision (TME) or non-operative management ("watch-and-wait") depending on response and clinical assessment.
  Interventions: Radiation: GTV 58.75 Gy/25 fractions(Simultaneous Integrated Boost); Drug: Concurrent Chemotherapy; Procedure: Total mesorectal excision (TME) surgery or non-operative management
- Control Arm (PGTV 50 Gy/25f) (Active Comparator): Radiotherapy: long course simultaneous integrated boost radiotherapy Gross tumor volume (GTV): A total dose of 50Gy delivered in 25 fractions using a simultaneous integrated boost approach.
  CTV: 45Gy/25f Mesorectum lymph node(GTVnd1):58.75Gy/25f Lateral lymph node（GTVnd2）：60Gy/25f Concurrent Chemotherapy: Concurrent administration of capecitabine (825 mg/m² twice daily, 5 days per week) or XELOX regimen during radiotherapy After treatment, patients will undergo restaging and proceed to total mesorectal excision (TME) or non-operative management ("watch-and-wait") depending on response and clinical assessment.
  Interventions: Radiation: GTV 50 Gy/25 fractions(Simultaneous Integrated Boost); Drug: Concurrent Chemotherapy; Procedure: Total mesorectal excision (TME) surgery or non-operative management

INTERVENTIONS:
Radiation: GTV 58.75 Gy/25 fractions(Simultaneous Integrated Boost) — Patients will receive neoadjuvant long course radiotherapy using VMAT or IMAT with daily image guided.
  Gross tumor volume (GTV): A total dose of 58.75Gy delivered in 25 fractions using a simultaneous integrated boost approach; CTV: 45Gy/25f; Mesorectum lymph node(GTVnd1):58.75Gy/25f ; Lateral lymph node（GTVnd2）：60Gy/25f;
  Arms: Experimental Arm (GTV 58.75 Gy/25f)
Radiation: GTV 50 Gy/25 fractions(Simultaneous Integrated Boost) — Patients will receive neoadjuvant radiotherapy with GTV 50 Gy in 25 fractions , delivered with IMRT or VMAT technique.
  CTV: 45Gy/25f; Mesorectum lymph node(GTVnd1):58.75Gy/25f; Lateral lymph node（GTVnd2）
  Arms: Control Arm (PGTV 50 Gy/25f)
Drug: Concurrent Chemotherapy — Concurrent administration of capecitabine (825 mg/m² twice daily, 5 days per week) or XELOX regimen during radiotherapy.
Procedure: Total mesorectal excision (TME) surgery or non-operative management — After treatment, patients will undergo restaging and proceed to total mesorectal excision (TME) or non-operative management ("watch-and-wait") depending on response and clinical assessment.

SUMMARY:
The goal of this clinical trial is to learn whether new adjuvant radiotherapy with gross tumor volume(GTV) escalated to 58.75 Gy can improve complete response (CR) rates compared with GTV dose of 50 Gy in adult patients (18-79 years) with locally advanced rectal adenocarcinoma (T3-T4/N+, M0) located ≤10 cm from the anal verge.The main questions it aims to answer are:

1. Does GTV simultaneously boost to 58.75 Gy/25f increase complete response (pCR or cCR) compared with 50 Gy/25f?
2. How do the two regimens differ in terms of progression-free survival (PFS), pelvic local control (LC), tumor regression grade (TRG), organ preservation, and treatment-related toxicity? Researchers will compare GTV 58.75 Gy/25f (experimental arm) versus GTV 50 Gy/25f (control arm) to see if dose escalation improves tumor response rate.

Participants will:

1. Receive neoadjuvant radiotherapy with one of the two PGTV dose escalated regimens (with concurrent chemotherapy: oral capecitabine or XELOX).
2. Undergo restaging with imaging and clinical assessment before surgery or observation.
3. Proceed to total mesorectal excision (TME), local excision, or "watch-and-wait" strategy depending on treatment response and patient preference.
4. Be followed regularly with clinical exams, imaging, endoscopy, and laboratory tests to assess efficacy, safety, and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and <80 years
2. Histologically confirmed rectal adenocarcinoma
3. Tumor located within 10 cm from the anal verge
4. MRI staging: T3-T4 and/or N+, M0 (AJCC 8th edition)
5. ECOG performance status 0-2
6. Adequate bone marrow function: WBC ≥3×10⁹/L, ANC ≥1.5×10⁹/L, PLT ≥100×10⁹/L, Hb ≥90 g/L
7. Adequate liver function: TBIL ≤1.5 × ULN, ALT/AST ≤2.5 × ULN
8. Adequate renal function: Cr ≤1.5 × ULN or CCr ≥60 mL/min
9. Signed informed consent

Exclusion Criteria:

1. Prior rectal cancer surgery
2. Prior induction chemotherapy, immunotherapy, or pelvic radiotherapy
3. History of other malignancies
4. History of chronic colitis, ulcerative colitis, or nonspecific proctitis
5. Pregnant or breastfeeding women
6. Active infection or fever
7. Severe uncontrolled comorbidities (e.g., unstable heart disease, renal disease, chronic hepatitis, uncontrolled diabetes, psychiatric disorders)
8. Inability to comply with study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
CR | 1 year
  primary tumor achieved pathological complete response or clinical complete response.

SECONDARY OUTCOMES:
3-year disease free suvival rate | 3 years
  The proportion of patients from the initiation of surgery to tumor recurrence or death within 3 years
3-year local control rate | 3 years
  The proportion of patients absence of pelvic tumor progression, including primary tumor regrowth or regional lymph node progression, within 3 years after randomization.
Tumor Regression Grade | 1 year
  Pathological tumor regression grade (TRG) according to CAP criteria.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 3 years
  Acute and late adverse events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Organ Preservation Rate | 1 year
  The proportion of patients who retain anal sphincter function without permanent stoma, including watch-and-wait, Dixon procedure or sphincter-preserving resection.